CLINICAL TRIAL: NCT05752292
Title: Optimizing a Scalable Intervention to Maximize Guideline-recommended Diabetes Testing After GDM
Brief Title: Study to Understand Risk Information to Support and Empower
Acronym: SUNRISE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1826240; R01DK122087 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-03-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetes, Gestational; Diabetes Mellitus, Type 2
Keywords: Gestational Diabetes; Diabetes Mellitus, Type 2 Prevention; Preventive Health Services; Health Communication
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Standard health message + VA + TRI + MI+ AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Tailored Risk Information (TRI); Behavioral: Motivational Interviewing-based (MI); Behavioral: Action planning (AP)
- Condition 2 (Experimental): Standard health message + VA + TRI + MI
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Tailored Risk Information (TRI); Behavioral: Motivational Interviewing-based (MI)
- Condition 3 (Experimental): Standard health message + VA + TRI + AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Tailored Risk Information (TRI); Behavioral: Action planning (AP)
- Condition 4 (Experimental): Standard health message + VA + TRI
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Tailored Risk Information (TRI)
- Condition 5 (Experimental): Standard health message + VA + MI+ AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Motivational Interviewing-based (MI); Behavioral: Action planning (AP)
- Condition 6 (Experimental): Standard health message + VA + MI
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Motivational Interviewing-based (MI)
- Condition 7 (Experimental): Standard health message + VA + AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA); Behavioral: Action planning (AP)
- Condition 8 (Experimental): Standard health message + VA
  Interventions: Behavioral: Standard Health Information; Behavioral: Values Affirmation (VA)
- Condition 9 (Experimental): Standard health message + TRI + MI+ AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Tailored Risk Information (TRI); Behavioral: Motivational Interviewing-based (MI); Behavioral: Action planning (AP)
- Condition 10 (Experimental): Standard health message + TRI + MI
  Interventions: Behavioral: Standard Health Information; Behavioral: Tailored Risk Information (TRI); Behavioral: Motivational Interviewing-based (MI)
- Condition 11 (Experimental): Standard health message + TRI + AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Tailored Risk Information (TRI); Behavioral: Action planning (AP)
- Condition 12 (Experimental): Standard health message + TRI
  Interventions: Behavioral: Standard Health Information; Behavioral: Tailored Risk Information (TRI)
- Condition 13 (Experimental): Standard health message + MI+ AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Motivational Interviewing-based (MI); Behavioral: Action planning (AP)
- Condition 14 (Experimental): Standard health message + MI
  Interventions: Behavioral: Standard Health Information; Behavioral: Motivational Interviewing-based (MI)
- Condition 15 (Experimental): Standard health message + AP
  Interventions: Behavioral: Standard Health Information; Behavioral: Action planning (AP)
- Condition 16 (Experimental): Standard health message
  Interventions: Behavioral: Standard Health Information

INTERVENTIONS:
Behavioral: Standard Health Information — Standard health information about postpartum screening and lifestyle programs for diabetes prevention
Behavioral: Values Affirmation (VA) — Interactive prompts to reflect on core personal values
  Arms: Condition 1; Condition 2; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Tailored Risk Information (TRI) — Interactive prompts to provide tailored information on risk factors for type 2 diabetes
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 2; Condition 3; Condition 4; Condition 9
Behavioral: Motivational Interviewing-based (MI) — Interactive prompts based on principles of motivational interviewing
  Arms: Condition 1; Condition 10; Condition 13; Condition 14; Condition 2; Condition 5; Condition 6; Condition 9
Behavioral: Action planning (AP) — Interactive prompts to problem solve challenges
  Arms: Condition 1; Condition 11; Condition 13; Condition 15; Condition 3; Condition 5; Condition 7; Condition 9

SUMMARY:
The aim of this trial is to test components of a digital health outreach intervention to promote uptake of postpartum screening and lifestyle programs for diabetes prevention among patients with gestational diabetes (GDM). The outreach intervention, designed to be interactive and delivered online, includes standard health information plus up to four theory-based components, targeting motivational and logistical barriers to engaging in diabetes preventive care during the postpartum period. The trial leverages the Multiphase Optimization Strategy (MOST) using a randomized factorial study design.

ELIGIBILITY:
Inclusion Criteria:

* Current pregnancy complicated by gestational diabetes mellitus (GDM)
* Age: 18 years and older
* Contact with the Kaiser Permanente Northern California (KPNC) Regional Perinatal Service Center
* Able to communicate in English

Exclusion Criteria:

* Diagnosis of diabetes before pregnancy
* Maternal or infant current hospitalization
* Pregnancy loss
* History of eating disorder
* Previously requested not to receive research invitations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Completion of recommended postpartum diabetes screening. | 4-12 weeks postpartum
  Completion of a 75-gram, 2-hour oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Completion of any recommended postpartum diabetes screening test. | 4-52 weeks postpartum
  Completion of any screening test (OGTT, fasting plasma glucose, or HbA1c)
Uptake of a lifestyle program for diabetes prevention. | 4-52 weeks postpartum
  Enrollment in a lifestyle program for diabetes prevention among women without type 2 diabetes mellitus according to any screening result

CONTACTS AND LOCATIONS:
Overall Officials: Susan D Brown, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Kaiser Permanente Northern California, Pleasanton, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT05752292/ICF_000.pdf